CLINICAL TRIAL: NCT05206123
Title: Sexual Health Needs of Adolescents Living With HIV Since Childhood : a Qualitative Study
Brief Title: Sexual Needs of Adolescents Living With HIV Since Childhood
Acronym: SSVIH
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP211568; 2021-A02820-41 (Other: ID-RCB)
Record Dates: First submitted 2021-12-20; First posted 2022-01-25 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Hiv; Perinatal HIV Infection
Keywords: HIV; sexual Health; adolescent; sexual needs
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents with perinatal acquired HIV infection: group of Adolescents with perinatal acquired HIV infection
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Patients will be interviewed with a semi-structured qualitative interview in order to know how they lived their first sexual experiences and their sex lives during their adolescence

SUMMARY:
To improve the knowdelge about the sexual health needs of perinatally HIV-infected adolescents living in France.

DETAILED DESCRIPTION:
20 individual semi-structured interviews will be conducted with 20 young adults living with HIV sinc childhood and living in France. The aim of this study is to identify their sexual needs through exploring their personal experience of sexuality during their adolescence. The investigator intend to explore communication about the disease and sexuality within their families ; communication about sexual health with health care professionnals ; whether sexuality has arrose difficulties related to their chronic condition such as rejection or sadness ; whether there are differences in sexual needs regarding gender. A thematic analysis will be conducted by three researchers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 25 yo
* HIV-1 or HIV-2 diagnosis before the age of 13
* non opposition to participate to the study
* be affiliated to a social security scheme (except Aide Médicale de l'Etat (AME))

Exclusion Criteria:

* having contracted HIV infection through sexual contact
* persons under guardianship or custodianship, or deprived of their liberty by a judicial or administrative decision
* associated illnesses or disabilities that makes participation impossible

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young adults with a perinatally acquired HIV infection
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Qualitative analysis | through study completion, an average of 1 year
  emerging themes describing the experience of their sexual health needs from the content analysis of the transcribed interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Maison de Solenn, Paris, France

IPD SHARING:
Plan to Share IPD: No